CLINICAL TRIAL: NCT03886129
Title: The Assessment of Cerebral Haemodynamics in Patients With Transient Ischaemic Attack: A Transcranial Doppler Study
Brief Title: Cerebral Haemodynamics in Transient Ischaemic Attack
Status: Terminated | Type: Observational
Why Stopped: COVID19 affected recruitment
Sponsor: University of Leicester (Other)
Responsible Party: Sponsor
Other Study IDs: 0694
Record Dates: First submitted 2019-03-20; First posted 2019-03-22 (Actual); Last update posted 2021-05-28 (Actual); Status verified 2021-05

CONDITIONS: Transient Ischemic Attack
MeSH Terms: conditions — Ischemic Attack, Transient | interventions — Ultrasonography, Doppler, Transcranial

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Participants with Transient Ischaemic Attack: Inclusion Criteria:
  * Willing to participate
  * Capacity to consent
  * Aged >18 years
  * Able (in the Investigator's opinion) and willing to comply with all study requirements
  * A diagnosis of acute (≤7 days) TIA, made by a specialist that fulfils the 2009 American Heart Association definition of TIA
  * Good understanding of written and verbal English
  Exclusion Criteria:
  * Unwilling to take part
  * Unable to consent
  * Aged <18 years
  * Unable (in the Investigator's opinion) or unwilling to comply with any study requirements
  * Female participants who are pregnant, lactating or planning pregnancy during the course of the study
  * Atrial fibrillation
  * Severe heart failure (Ejection Fraction <30%)
  * Severe respiratory disease
  * Inadequate bilateral transcranial Doppler windows
  * Carotid stenosis ≥70% (unilateral or bilateral)
  * Participant enrolled in an interventional research study.
  * Poor understanding of written and verbal English
  Interventions: Diagnostic Test: Transcranial Doppler Ultrasound (TCD)
- Healthy Control Participants: Inclusion Criteria:
  * Willing to participate
  * Capacity to consent to the study
  * Aged >18 years
  * Able (in the Investigator's opinion) and willing to comply with all study requirements
  * Good understanding of written and verbal English
  Exclusion Criteria:
  * Unwilling to take part
  * Unable to consent
  * Aged <18 years
  * Unable (in the Investigator's opinion) or unwilling to comply with any study requirements
  * Female participants who are pregnant, lactating or planning pregnancy during the course of the study
  * Atrial fibrillation
  * Severe heart failure (Ejection Fraction <30%)
  * Severe respiratory disease
  * Inadequate bilateral transcranial Doppler windows
  * Carotid stenosis ≥70% (unilateral or bilateral)
  * Participant enrolled in an interventional research study.
  * Poor understanding of written and verbal English
  Interventions: Diagnostic Test: Transcranial Doppler Ultrasound (TCD)

INTERVENTIONS:
Diagnostic Test: Transcranial Doppler Ultrasound (TCD) — Participants will undergo an assessment of brain blood flow using TCD, with two small ultrasound probes held in place on the temples with a customised headframe. During the assessment, heart rate, breathing and blood pressure will also be monitored using a 3 lead ECG, nasal capnography and Finometer® respectively. The assessment will comprise three recordings. Firstly, participants will sit quietly for 5 minutes. Next, they will be asked to sit quietly for one minute before standing and remaining standing for 5 minutes. Lastly, they will be asked to stand and then complete a squat-stand manoeuvre in time with a computer sequence. A tilt sensor attached to the thigh will measure the efficiency and angle of the squatting motion. The squat-stand manoeuvre will consist of 15 squats and participants will be informed that they should try and complete all 15 squats if possible.

SUMMARY:
Adequate brain blood flow is essential for brain survival and function. Brain blood flow is kept relatively constant by a process called cerebral autoregulation (CA). CA is impaired in various diseases including head injury, diabetes, Alzheimer's, pre-eclampsia and stroke. In stroke, impaired CA is associated with poor outcomes. A transient ischaemic attack (TIA) is the same as a stroke, except the symptoms only last for a short amount of time and resolve spontaneously. TIAs are sometimes called mini-strokes and are a major warning sign of strokes. There have been lots of studies of CA in stroke, but very few studies of CA in TIA. Brain blood flow and CA can be studied non-invasively with Transcranial Doppler ultrasound (TCD).

Study aim: To investigate whether CA is impaired in patients with TIA

20 patients with acute TIA (within 7 days), and 20 healthy controls will be recruited from the specialist TIA clinic at University Hospitals of Leicester NHS Trust. Participants will be eligible if they are aged over 18 and can consent to participate. They won't be able to participate if they have severe heart failure, an irregular heartbeat, blocked neck blood vessels, severe breathing problems, or if they are pregnant.

Participants will undergo an assessment of brain blood flow using TCD, during which their heart rate, breathing and blood pressure will also be monitored. During the assessment participants will sit quietly before being asked to stand and then complete a squat-stand manoeuvre in time with a computer sequence. The research visit will take approximately 90 minutes, the assessment itself will take approximately 1 hour and participants only need to attend once.

DETAILED DESCRIPTION:
Adequate brain blood flow is essential for brain survival and function. Brain blood flow is kept relatively constant by a process called cerebral autoregulation (CA). CA is impaired in various diseases including head injury, diabetes, Alzheimer's dementia, pre-eclampsia and stroke. In stroke, impaired CA is associated with early deterioration and the need for emergency surgery to relieve brain swelling. Impaired CA in stroke has also been shown to be related to stroke severity and functional outcomes.

A transient ischaemic attack (TIA), also known as a mini-stroke, is the same as a stroke, except that the symptoms only last for a short amount of time and resolve spontaneously. Every year at least 46,000 people in the United Kingdom have a TIA for the first time. TIA is strongly predictive of future stroke, and the risk is heavily front loaded; one in 12 people will have a full stroke within a week of having a TIA. Prompt assessment following a TIA helps to reduce this risk. Indeed, urgently investigating and treating people who have a TIA in a specialist clinic reduces their risk of another stroke by 80%. However, some people will unfortunately go on to have a stroke despite this, and the reasons for this are not always clear. Furthermore, although TIAs fully resolve, around 70% of people report long term effects after a TIA including memory loss, tiredness and low mood.

Brain blood flow and CA can be studied using ultrasound which is passed through the skull, known as Transcranial Doppler ultrasonography (or TCD). Ultrasound has been tried and tested over many years and unlike CT or MRI scans, does not use any radiation. It is also inexpensive, and can be used in patients with pacemakers.

In order to study CA, it is necessary to see what happens to brain blood flow when there are changes in blood pressure. Although some people have natural ups and downs in their blood pressure at rest, these are not always big enough to study brain blood flow effectively. Larger changes in blood pressure can be induced with challenges such as placing hands in ice cold water, or inflating large blood pressure cuffs on the tops of the legs before suddenly releasing them. These can be uncomfortable for participants. More recently, squat-stand manoeuvres (SSMs) have also been shown to produce large changes in blood pressure. They have been shown to be safe and well tolerated in various populations including heart transplant recipients, young and old healthy controls, and patients with Alzheimer's dementia. It has recently been shown that reliable CA data can be obtained from as few as three SSMs.

There have been lots of studies of CA in stroke, but very few studies of CA in TIA. The small studies that are available are conflicting about whether brain blood flow and CA are altered in TIA. The aim of this study is therefore to investigate whether CA is impaired in patients with TIA. If CA is impaired in patients with TIA, then it may be possible to identify abnormalities in brain blood flow that can help predict who might go on to suffer a stroke, or suffer other complications.

This is a single-centre, case-control study being undertaken at the University Hospitals of Leicester NHS Trust.

Once ethical approvals, and all relevant sponsorship and regulatory approvals, are in place 20 patients with acute TIA (within 7 days of event), and 20 healthy controls will be recruited from the specialist TIA clinic at University Hospitals of Leicester NHS Trust. Medical records will be reviewed by the direct care team to ensure participants meet the inclusion and exclusion criteria. Participants will be eligible if they are aged over 18 and can consent to participate. They won't be able to participate if they have severe heart failure, an irregular heartbeat, blocked neck blood vessels, severe breathing problems, or if they are pregnant. Eligibility screening will only be undertaken by the direct clinical care team for potential participants. Participants will be approached at their clinical consultation in the specialist TIA clinic by consultants, registrars or specialist nurses to determine study interest prior to referral to the researcher and provision of study specific information. A poster advertising the study will be displayed in the TIA clinic waiting room. Both participants with TIA, and healthy controls (those without a diagnosis of TIA) will be recruited from the clinic. Healthy spouses, friends or partners of patients with TIA will be asked if they would like to participate in the study as a healthy control subject.

Participants who meet the inclusion criteria will attend the Leicester Cerebral Haemodynamics in Ageing and Stroke Medicine (CHiASM) research laboratory. Formal, written consent will be obtained, followed by an ultrasound check of their brain blood flow. In approximately 5-37% of patients we are not able to perform the ultrasound procedure as the blood vessels cannot be seen through the skull, which would prevent them from enrolling into the study. Following this, background information on age, sex, medical conditions, and medication use will be collected. The Edinburgh handedness inventory will be completed to determine left or right hand dominance, and the office of National Statistics questionnaire to determine ethnicity.

Participants will then undergo an assessment of brain blood flow using TCD, with two small ultrasound probes held in place on the temples with a customised headframe. During the assessment, heart rate, breathing and blood pressure will also be monitored. Heart rate will be monitored using a 3 lead ECG, blood pressure will be monitored using a cuff on the finger with the arm supported in a sling, and breathing will be monitored using nasal tubes. The assessment will consist of three recordings. Firstly, participants will sit quietly for 5 minutes. Next, they will be asked to sit quietly for one minute before standing and remaining standing for 5 minutes. Lastly, they will be asked to stand and then complete a squat-stand manoeuvre in time with a computer sequence. A tilt sensor will be attached to the thigh to measure the efficiency and angle of the squatting motion. The squat-stand manoeuvre will consist of 15 squats and participants will be informed that they should try and complete all 15 squats if possible. However, if they wish to stop before this, they should make the investigator aware during a standing period and remain standing for 90 seconds before the equipment is disconnected.

The research visit will take approximately 90 minutes, the assessment itself will take approximately 1 hour and participants only need to attend once.

ELIGIBILITY:
INCLUSION CRITERIA:

HEALTHY CONTROLS:

* Willing to participate
* Capacity to consent to the study
* Aged over 18 years
* Able (in the Investigator's opinion) and willing to comply with all study requirements
* Good understanding of written and verbal English

TIA PATIENTS:

* Willing to participate
* Capacity to consent to the study
* Aged over 18 years
* Able (in the Investigator's opinion) and willing to comply with all study requirements
* A diagnosis of acute (≤7 days) TIA, made by a specialist in the TIA clinic at University Hospitals of Leicester NHS Trust that fulfils the 2009 American Heart Association definition of TIA
* Good understanding of written and verbal English

EXCLUSION CRITERIA:

ALL PARTICIPANTS (HEALTHY CONTROLS AND TIA PATIENTS)

* Unwilling to take part
* Unable to consent
* Aged under 18 years
* Unable (in the Investigator's opinion) or unwilling to comply with any study requirements
* Female participants who are pregnant, lactating or planning pregnancy during the course of the study
* A diagnosis of atrial fibrillation
* A diagnosis of severe heart failure (Ejection Fraction <30%)
* Severe respiratory disease
* Inadequate bilateral transcranial Doppler windows (see section 8.3)
* Carotid stenosis ≥70% (unilateral or bilateral)
* Participant enrolled in an interventional research study.
* Poor understanding of written and verbal English

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 20 adult patients with acute TIA (within 7 days), and 20 healthy controls will be recruited from the specialist TIA clinic at University Hospitals of Leicester NHS Trust.
Sampling Method: Non-Probability Sample
Enrollment: 2 (Actual)
Dates: Start 2019-04-16 (Actual); Primary Completion 2021-03-31 (Actual); Study Completion 2021-03-31 (Actual)

PRIMARY OUTCOMES:
Beat-to-beat brain blood flow velocity | 6 months
  To determine the beat-to-beat brain blood flow velocity of both TIA and Healthy Control (HC) subjects during performance of a squat-stand manoeuvre.

SECONDARY OUTCOMES:
Autoregulation index | 6 months
  To determine other beat-to-beat brain blood flow parameters, specifically autoregulation index (ARI), of both TIA and HC subjects during performance of a squat-stand manoeuvre.

CONTACTS AND LOCATIONS:
Overall Officials: Thompson G Robinson, MD, Principal Investigator — University of Leicester
Locations (1):
- University Hospitals of Leicester NHS Trust, Leicester, United Kingdom

IPD SHARING:
Plan to Share IPD: No
There is no plan to make individual participant data (IPD) available to other researchers.
  Anonymised cohort data may be shared with researchers from other Departments or Universities conducting similar research. Explicit written consent for the sharing of such data will be obtained from participants.

DOCUMENTS (3):
  • Study Protocol and Statistical Analysis Plan (2019-02-20): https://cdn.clinicaltrials.gov/large-docs/29/NCT03886129/Prot_SAP_000.pdf
  • Informed Consent Form: Healthy Control Participants (2019-02-20): https://cdn.clinicaltrials.gov/large-docs/29/NCT03886129/ICF_001.pdf
  • Informed Consent Form: TIA Participants (2019-02-20): https://cdn.clinicaltrials.gov/large-docs/29/NCT03886129/ICF_002.pdf